CLINICAL TRIAL: NCT03270761
Title: A Multi-center Study on Iridocorneal Endothelial (ICE) Syndrome in China
Brief Title: Zhongshan Iridocorneal Endothelial Syndrome Study (ICEs)
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: ICE study group (Unknown)
Responsible Party: Principal Investigator, Xiulan Zhang, MD,PhD, Sun Yat-sen University
Other Study IDs: 2017KYPJ071
Record Dates: First submitted 2017-08-24; First posted 2017-09-01 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 12ml Blood will be collected. Aqueous humor，iris,or excised corneal will be gathered if trabeculectomy,drainage shunt valve implantation, or penetrating keratoplasty needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
This is a multi-center study to report the demographic profile, clinical features, and management in patients with Iridocorneal endothelial (ICE) syndrome in China.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ICE syndrome;
* Those willing to sign the informed consent.

Exclusion Criteria:

* Patients who don't sign the informed consent or abide by the study procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICE syndrome patients identified and enrolled from 50 study centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Management in patients with Iridocorneal endothelial (ICE) syndrome | through study completion, an average of 1 year
  Record the number of medication treating corneal edema or glaucoma, and surgery (anti-glaucoma surgery, keratoplasty)

SECONDARY OUTCOMES:
Demographic profile of patients | 1 day
  Range of age, gender

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD,PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No